CLINICAL TRIAL: NCT06422364
Title: Assessment of the Safety and Efficacy of Weighted Wearable Blankets in Healthy Infants During Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: External to study controversy has arisen around safety of the product. Due to concerns raised by USCPSC and the AAP, the PI has terminated site participation.
Sponsor: Indiana University (Other)
Collaborators: Dreamland Baby Co. (Unknown)
Responsible Party: Principal Investigator, Harish Rao, Assistant Professor of Clinical Pediatrics, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21638
Record Dates: First submitted 2024-04-26; First posted 2024-05-21 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Sleep
Keywords: Sleep; Healthy; Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Nap Polysomnogram (Experimental): All healthy infants under 3 months of age that met inclusion criteria were assigned to complete a nap polysomnogram while wearing a weighted wearable blanket provided by Dreamland Baby Co.
  Interventions: Device: Weighted Wearable Blanket provided by Dreamland Baby Co.
- Overnight Polysomnogram (Experimental): All healthy infants over 3 months of age that met inclusion criteria were assigned to complete an overnight polysomnogram while wearing a weighted wearable blanket provided by Dreamland Baby Co.
  Interventions: Device: Weighted Wearable Blanket provided by Dreamland Baby Co.

INTERVENTIONS:
Device: Weighted Wearable Blanket provided by Dreamland Baby Co. — All infants will be placed in a weighted wearable blanket, provided by Dreamland Baby Co., and complete a nap polysomnogram.
  Arms: Nap Polysomnogram
Device: Weighted Wearable Blanket provided by Dreamland Baby Co. — All infants will be placed in a weighted wearable blanket, provided by Dreamland Baby Co., and complete an overnight polysomnogram.
  Arms: Overnight Polysomnogram

SUMMARY:
The goal of this clinical trial is to assess the risk of an infant overheating and/or experiencing lowered respiration via measurement of vital signs in a controlled clinical environment while wearing a weighted wearable blanket in male/female infant healthy volunteers, 0-12 months of age.

The main questions it aims to answer are:

Primary Objective: To pilot an investigation on the impact of weighted wearable blankets on vital signs and infant movement in healthy infants during nap polysomnogram.

Secondary Objective: To investigate the efficacy of weighted wearable blankets on sleep patterns in healthy infants during overnight sleep.

DETAILED DESCRIPTION:
To date, there is no evaluation of the safety or efficacy of weighted wearable blankets on healthy infants during overnight use in the peer-reviewed scientific literature. These are the conditions in which these products are used by consumers, with infants sleeping unobserved throughout the night. Given the rising popularity in the use of weighted wearable blankets in infants and the risk speculated, a study of the potential impact of weighted wearable blankets on infant vital signs is warranted.

Study Design: Direct observational pilot study of the safety of weighted wearable blankets on a minimum (10) healthy infants aged 0-12 months with nap polysomnogram. Participants will be placed in a weighted wearable blanket, in accordance with their age/weight/height, by their parent or caregiver under the supervision of a member of the study team. After being put to sleep on their back, the participant will remain in the weighted wearable blanket until completion of the nap polysomnogram.

There are stopping parameters (outlined elsewhere) that will be used for this study. If any of the stopping parameters are met, the weighted blanket will be opened to assess if the weighted blanket is responsible for the change. If determined yes, the weighted blanket will be removed and the nap polysomnogram will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Ability of parent, caregiver or legal guardian/representative to understand a written informed consent document and choose to participate in the study
* 0-12 months of age
* Weight greater than or equal to 8 pounds
* Gestational age 37 weeks or greater
* Health status: healthy infant without underlying cardiac, neurological, or pulmonary disorders
* Infant is naive to a weighted wearable blanket

Exclusion Criteria:

* Health status: medical diagnosis associated with underlying cardiac, neurological, or pulmonary disorder
* Weight < 8 pounds
* Gestational age < 37 weeks
* Gestational use of marijuana, alcohol, or illicit drugs
* Home environment: use of cigarettes, vaping, e-cigarettes, or marijuana
* Infant is not naive to a weighted wearable blanket

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Rao, MD, Principal Investigator — Riley Hospital for Children at Indiana University Health
Locations (1):
- Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Dreamland Baby website utilized a link for potential participants to express their interest in the study. A member of the study team made contact by email and then telephone to conduct a recruitment/screening questionnaire. A nap polysomnogram was scheduled during daytime hours for participants that met inclusion criteria and were under 3 months of age. Infants that met inclusion criteria and were greater than 3 months of age were scheduled for an overnight polysomnogram.
Pre-assignment Details: 6 enrolled participants met inclusion criteria; 4 enrolled participants completed the nap polysomnogram; 2 enrolled participants were withdrawn due to study closure prior to scheduled overnight polysomnogram dates. Those that completed the nap polysomnogram also completed a one-week post survey.
Period: Overall Study
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Started | 4 | 2
Completed | 4 | 0
Not Completed | 0 | 2
Not completed — Withdrawn due to study closure | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: days] — Age at Time of Informed Consent
  days | 59 (14.118545723032) | 114.5 (23.334523779156) | 77.5 (32.402160421799)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Heart Rate
Description: Measured by EKG
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
beats per minute | 122 (18.98) |

2. Primary Outcome: Average Respiratory Rate
Description: Measured by Respiratory effort belts
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
respirations per minute | 42.25 (8.42) |

3. Primary Outcome: Average Body Temperature
Description: Manually measured by ear thermometer
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Mean (Standard Deviation); unit: average body temperature, Celsius
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
average body temperature, Celsius | 36.95 (0.13) |

4. Primary Outcome: Average Oxygen Saturation
Description: Measured by pulse oximetry
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Mean (Standard Deviation); unit: oxygen saturation percentage
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
oxygen saturation percentage | 97.25 (0.5) |

5. Primary Outcome: Number of Infants With Observed Head Movement
Description: The clinical technician will be asked to report any observed infant movements during the polysomnogram. The technician will report either Yes or No to this question.
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Count of Participants; unit: Participants
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
Participants | 4 |

6. Primary Outcome: Number of Infants With Observed Arm Movement
Description: as for outcome 5
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Count of Participants; unit: Participants
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
Participants | 1 |

7. Primary Outcome: Number of Infants With Observed Body Movement
Description: as for outcome 5
Time Frame: Day 1, during polysomnogram, up to 8 hours
Population: The study was closed before participants could complete the overnight polysomnogram.
Measure: Count of Participants; unit: Participants
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
Number analyzed (Participants) | 4 | 0
Participants | 4 |

8. Secondary Outcome: Efficacy of Weighted Wearable Blankets on Sleep Patterns in Healthy Infants During Overnight Sleep
Description: The study was closed before any overnight studies were completed; therefore, no data for this objective was collected.
Time Frame: Day 1, during polysomnogram, up to 12 hours
Population: No overnight studies were completed; therefore, no data for this objective was collected.
Arm/Group | Overnight Polysomnogram
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected after informed consent was signed until the one-week post survey was completed. The maximum amount of time participants spent in the study was 37 days, which included signing the informed consent, completing the nap polysomnogram and completing the one-week post survey.
Description: On the one-week post survey, parents were asked if their child had experienced any changes in their baseline health. If parent response was yes, parent was invited to describe what was experienced. A staff member then interviewed parent to collect adverse event information.
Arm/Group | Nap Polysomnogram | Overnight Polysomnogram
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nap Polysomnogram (N=4) | Overnight Polysomnogram (N=2)
Left Eye Discharge (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT06422364/Prot_SAP_000.pdf